CLINICAL TRIAL: NCT06867679
Title: Effects of Recreational Soccer Training on Physical Fitness and Gross Motor Coordination in Prepubertal Boys and Girls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/G-III/RCR&AHS/B42-177
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy Male and Female Subjects
Keywords: Physical Fitness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recreational Soccer Training (Boys Group) (Experimental): Prepubertal Girls Group
  Interventions: Other: Recreational Soccer Training (Boys Group)
- Recreational Soccer Training (Girls Group) (Experimental): Prepubertal Girls Group
  Interventions: Other: Recreational Soccer Training (Girls Group)

INTERVENTIONS:
Other: Recreational Soccer Training (Boys Group) — This group will have 3 training sessions per week, with each session lasting 60 minutes (13). The session will include: Warm-up (10 minutes): Light jogging, Dynamic stretching (Arm circles, Leg swings, Hip circles), Mobility exercises (Ankle roll, Trunk rotations),Technical Skills Training (20 minutes):Dribbling, passing, and shooting drills, Small-Sided Games (20 minutes): 3v3 or 4v4 games emphasizing teamwork, passing, and movement off the ball.Cool Down (10 minutes):Light jogging, Static stretching, Breathing exercises. Training Progression: Weeks 1-2: Basic skills and small-sided games, Weeks 3-5: Increased drill complexity, Weeks 6-8: Enhanced tactical awareness and structured gameplay.
  Other Names: Prepubertal Boys Group
  Arms: Recreational Soccer Training (Boys Group)
Other: Recreational Soccer Training (Girls Group) — This group will have 3 training sessions per week, with each session lasting 60 minutes (13). The session will include: Warm-up (10 minutes): Light jogging, Dynamic stretching (Arm circles, Leg swings, Hip circles), Mobility exercises (Ankle roll, Trunk rotations),Technical Skills Training (20 minutes):Dribbling, passing, and shooting drills, Small-Sided Games (20 minutes): 3v3 or 4v4 games emphasizing teamwork, passing, and movement off the ball.Cool Down (10 minutes):Light jogging, Static stretching, Breathing exercises. Training Progression: Weeks 1-2: Basic skills and small-sided games, Weeks 3-5: Increased drill complexity, Weeks 6-8: Enhanced tactical awareness and structured gameplay.
  Other Names: Prepubertal Girls Group
  Arms: Recreational Soccer Training (Girls Group)

SUMMARY:
Physical activity is essential for the healthy development of children, contributing significantly to their physical fitness and motor skills. Prepubertal children experience changes in physical growth. During the prepubertal phase, engaging in regular physical activity can lead to substantial improvements in cardiovascular health, muscular strength, agility, and coordination. Physical fitness has been recognized as a key determinant in healthy lifestyles based increasingly on criteria referenced to general health. However, many children and adolescents are only exposed to vigorous physical activity during school based physical education classes. That way, schools seem to provide an excellent setting to enhance physical activity and physical fitness levels. Soccer, a widely popular sport, offers an engaging and enjoyable way for children to improve their physical fitness and gross motor coordination.

This study aims to investigate the effects of recreational soccer training on physical fitness and gross motor coordination in prepubertal boys and girls and to compare the effects of recreational soccer training between boys and girls. This current study will be a clinical trial; data will be calculated from Dar-e-Arqam School, upper mall Lahore. A total of 70 prepubertal children (35 boys and 35 girls) will be recruited for this study. Inclusion criteria for the study will be 7 to 9 years old boys and girls. participants should be in good general health, without any medical condition that could affect their ability to participate in physical activities. Individuals with physical disabilities or impairments that prevent them from engaging in soccer activities will be excluded. Participants will be divided into two experimental groups: Group A (boys) and Group B (girls). Both groups will undergo the same soccer training program. The soccer training program will consist of sessions held thrice a week for 8 weeks, each lasting 60 minutes.Outcomes to be analyzed will be Physical fitness and Gross motor coordination. Data collection will be done before and after the intervention. Tools used for data collection will be Physical fitness test battery for children to assess physical fitness and rohrer's index will be used to assess somatotype. Gross motor coordination will be evaluated using the Körperkoordinations test für Kinder (KTK) test battery. Data will be analyzed through SPSS version 26.00.

ELIGIBILITY:
Inclusion Criteria:

* Children between age 7 to9
* Flamingo balance test between 11-14
* Both genders

Exclusion Criteria:

* Presence of any chronic medical condition
* Children who areinvolved inother training program
* Having any physical disability or impairment

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Physical Fitness Test Battery for Children | Baseline and 8th Week
  Physical fitness test battery for children has been found to be highly reliable tool with interclass correlation coefficients for individual test items and total score ranging from .54 to .92
Körperkoordinationstest für kinder (KTK) for Gross Motor Coordination | Baseline and 8th Week
  The Körperkoordinationstest für Kinder (KTK) is a widely used test to assess motor coordination in children. KTK has high test-retest reliability ranging from o.80 to 0.96, indicating that children's performance on the test is consistent over repeated administrations. The test involves components of Motor Coordination, such as balance, rhythm, strength, laterality, speed, and agility.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- CDGL Boys High School, Upper Mall, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammami M, Negra Y, Billaut F, Hermassi S, Shephard RJ, Chelly MS. Effects of Lower-Limb Strength Training on Agility, Repeated Sprinting With Changes of Direction, Leg Peak Power, and Neuromuscular Adaptations of Soccer Players. J Strength Cond Res. 2018 Jan;32(1):37-47. doi: 10.1519/JSC.0000000000001813. PMID 28678768